CLINICAL TRIAL: NCT02515344
Title: Impact of the Distribution to Attending Physicians of a Nominative List of Their Patients Not Participating in the Organised Screening of Colorectal Cancer: Randomised Study Measuring the Impact on Participation
Brief Title: Impact of the Distribution to Attending Physicians of a Nominative List of Their Patients Not Participating in the Organised Screening of Colorectal Cancer
Acronym: IDLN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Public Health Insurance (Unknown); Université de Nantes (Other); Organisms in charge of local cancer screening programs - France (Unknown); Local Cancer Registry - France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC12_0497
Record Dates: First submitted 2015-07-21; First posted 2015-08-04 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: Patients; early detection of cancer; patient compliance
MeSH Terms: conditions — Colorectal Neoplasms; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: nominative list (Experimental): Providing a list of patients not compliant with CRC sreening
  General Practitioners allocated to the intervention group (A) will receive:
  * a nominative list of their patients who were not compliant to colorectal cancer screening.
  * a document providing general information about colorectal cancer screening
  Interventions: Other: Providing a list of patients not compliant with CRC sreening; Other: Providing general information about CRC sreening
- B: general information (Active Comparator): Providing general information about CRC screening
  General Practitioners allocated to group (B) will receive:
  - a document providing general information about colorectal cancer screening (but will not receive the nominative list of patients non compliant to colorectal cancer screening)
  Interventions: Other: Providing general information about CRC sreening
- C: usual practice (No Intervention): General Practitioners allocated to group (C) will not receive any information (as in usual practice)

INTERVENTIONS:
Other: Providing a list of patients not compliant with CRC sreening — GPs allocated to the intervention group (A) will receive a list of the patients who are not compliant to colorectal cancer screening, while GPs allocated to the others groups will not receive this information.
  Arms: A: nominative list
Other: Providing general information about CRC sreening
  Arms: A: nominative list; B: general information

SUMMARY:
Objective : to demonstrate that providing to GPs a list of their patients who are not compliant to colorectal cancer screening will 1) enhance patient participation to screening, and 2) decrease the proportion of cancer diagnosed outside the screening organisation. Design : Randomised controlled study, 3 parallel arms. Enrollment: GPs allocated in the 3 groups of the study will be all GPs 1) from the "Loire-Atlantique and Vendée" geographic area (1300 GPs on average) and 2) who have more than 100 patients in their patient list (based on data provided by the Healthcare Insurance System Services). Patients will be eligible to the study depending on their eligibility to the Faecal Occult Blood Test for colorectal cancer screening : 1) they should be older than 50 and younger than 74; 2) they should not have a personal history of colorectal cancer (or history of adenoma bigger than 1 cm) nor a family history of colorectal cancer. Main outcomes measures : Patient participation to colorectal cancer screening, and number of cancers screened in (versus diagnosed outside) the screening procedure.

DETAILED DESCRIPTION:
Background:

Participation rate for colorectal cancer screening in France is 39%. In a Cochrane review, patient participation rates to colorectal cancer screening varies from 30 to 60%. Policy makers usually consider that these participation rates should be higher, based on the premise that the impact of the screening mainly depends on patient participation. In France, patients at average risk of colorectal cancer are eligible to the Faecal Occult Blood Test for colorectal cancer screening if: 1) they are older than 50 and younger than 74; 2) they have no personal history of colorectal cancer (or history of adenoma bigger than 1 cm) and no family history of colorectal cancer.

Objective:

To demonstrate that providing to GPs a list of their patients who are not compliant to colorectal cancer screening will 1) enhance patient participation to screening, and 2) decrease the proportion of cancer diagnosed outside the screening organisation. Design : Randomised controlled study, 3 parallel arms.

Design:

Randomized controlled study. 3 parallel arms.

Setting:

Primary care setting in France.

Enrollment:

In this study, the intervention will focus on the GP. The statistical unit for the results analysis will be the GP. GPs allocated in the 3 groups of the study will be all GPs 1) from the "Loire-Atlantique and Vendée" geographic area (1300 GPs on average) and 2) who have more than 100 patients in their patient list (based on data provided by the Healthcare Insurance System Services).

Intervention:

GPs allocated to the intervention group (A) will receive a list of the patients who are not compliant to colorectal cancer screening, while GPs allocated to the others groups will not receive the corresponding information.

Randomization:

3 groups : (A) GPs will receive a list of the patients who are not compliant to colorectal cancer screening, (B) GPs will receive a document providing general information on colorectal cancer screening, (C) GPs will not receive any specific document (they continue regular practice).

Primary outcome measure: Patient participation to colorectal cancer screening Secondary Outcome Measures: number of cancers screened in (versus diagnosed outside) the screening procedure.

ELIGIBILITY:
In this study, the statistical unit is the GP.

Inclusion Criteria:

GPs allocated in the 3 groups of the study will be all GPs

* 1) from the "Loire-Atlantique and Vendée" geographic area (1300 GPs on average)
* 2) who have more than 100 patients in their patient list (based on data provided by the Healthcare Insurance System Services).

Exclusion Criteria:

* GPs who have less than 100 patients in their patient list

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48649 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Patient participation rate to colorectal cancer screening | 12 months after starting date of the study

SECONDARY OUTCOMES:
Number of cancers screened in (versus diagnosed outside) the screening procedure. | 12 months after starting date of the study

REFERENCES:
- [Derived] Rat C, Pogu C, Le Donne D, Latour C, Bianco G, Nanin F, Cowppli-Bony A, Gaultier A, Nguyen JM. Effect of Physician Notification Regarding Nonadherence to Colorectal Cancer Screening on Patient Participation in Fecal Immunochemical Test Cancer Screening: A Randomized Clinical Trial. JAMA. 2017 Sep 5;318(9):816-824. doi: 10.1001/jama.2017.11387. PMID 28873160